CLINICAL TRIAL: NCT03027973
Title: Quality of Life Outcomes for Ulipristal Acetate and Tranexamic Acid in the Management of Heavy Menstrual Bleeding: A Pilot Randomized Control Trial
Brief Title: Quality of Life Outcomes for Ulipristal Acetate and Tranexamic Acid in the Management of Heavy Menstrual Bleeding
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI made the decision to not continue the study. It was at the Health Canada review stage.
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Almereau Prollius, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBLL07230904; 16-155 (Other: University of Saskatchewan Biomedical Research Ethics Board)
Record Dates: First submitted 2017-01-15; First posted 2017-01-23 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — ulipristal acetate; Tea; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPA Treatment Group (Experimental): UPA 5mg capsule daily + Placebo 2 capsules 4 times a day
  Interventions: Drug: UPA; Drug: Placebo (for TEA)
- TEA Treatment Group (Active Comparator): TEA 500mg 2 capsules 4 times a day + Placebo 1 capsule daily
  Interventions: Drug: TEA; Drug: Placebo (for UPA)

INTERVENTIONS:
Drug: UPA — Experimental drug
  Other Names: Ulipristal Acetate
  Arms: UPA Treatment Group
Drug: TEA — Active comparator
  Other Names: Tranexamic Acid
  Arms: TEA Treatment Group
Drug: Placebo (for UPA) — Sugar pill manufactured to mimic UPA 5 mg
  Arms: TEA Treatment Group
Drug: Placebo (for TEA) — Sugar pill manufactured to mimic TEA 500mg
  Arms: UPA Treatment Group

SUMMARY:
This study compares two treatments for the management of heavy menstrual bleeding, ulipristal acetate (UPA) and tranexamic acid (TEA), on health-related quality of life. Half of the participants will receive UPA and a placebo, and the other half will receive TEA and a placebo.

DETAILED DESCRIPTION:
UPA is approved by Health Canada for the treatment of signs and symptoms of uterine fibroids in adult women of reproductive age who are eligible for surgery. UPA is considered investigational for this study, as it has not been approved by Health Canada for the treatment of heavy menstrual bleeding in women who do not have uterine fibroids.

TEA is approved by Health Canada for prevention or reduction of bleeding in different conditions, including heavy periods. This treatment is available as part of routine care for regular heavy menstrual bleeding and is being used as the comparison treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are female and have a uterus
* Participants are between the ages of 18 and 51 years at the time of consent
* Participants have heavy menstrual bleeding as evidenced by their symptoms of subjective increased bleeding volume and desire to seek treatment
* The symptom of heavy menstrual bleeding has been present for most of the last 6 months
* Participants have regular menstrual cycles between 24 -38 days in length

Exclusion Criteria:

* Participants who are pregnant or have a positive urine β-hCG
* Participants whose bleeding is coming from a cervical, vaginal, urinary or gastrointestinal source
* Participants who are found to have or who have a previous diagnosis of uterine or cervical polyps, adenomyosis, or leiomyomas (fibroids)
* Participants who are found to have or who have had endometrial hyperplasia, cervical dysplasia or malignancy of any of the vulva, cervix, endometrium, breast or ovaries.
* Participants who have ovulatory dysfunction as defined by menstrual cycles that are irregular in frequency and regularity and are often punctuated with periods of amenorrhea
* Participants who are found to have or who have been diagnosed with a coagulopathy
* Participants who have a current genitourinary infection
* Participants who are desirous of becoming pregnant within the next four months
* Participants who have untreated or inadequately treated thyroid disease
* Participants who have a contraindication to either treatment including hypersensitivity
* Participants who are breastfeeding
* Participants with mild, moderate or severe hepatic impairment
* Participants with moderate or severe renal impairment
* Participants with severe asthma not controlled with oral glucocorticoids
* Participants with active disease, or history of deep vein thrombosis (DVT), pulmonary embolism (PE), cerebral thrombosis or with family history of thromboembolic disease
* Patients with subarachnoid hemorrhage
* Patients with acquired disturbances of colour vision
* Participants who are already on hormone based treatment including, progesterone only pills, combined oral contraceptive pill (COCP), Intrauterine System (IUS)

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Menorrhagia Multi-attribute Scale (MMAS) at 3 Months | At Baseline and repeated 3 months later
  The MMAS measures the impact of menorrhagia on health related quality of life (QoL) in six domains.

SECONDARY OUTCOMES:
Number of adverse events that occur | From Baseline visit to end of study 3 months later
  The subjective change in symptoms will be assessed based on recordings in the study diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Almereau Prollius, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon Obstetric and Gynecologic Consultants, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No